CLINICAL TRIAL: NCT04232202
Title: Post-extraction Treatment With Er:YAG and Nd:YAG Lasers - Socket Preservation
Brief Title: Socket Preservation With Er:YAG and Nd:YAG Lasers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krizaj d.o.o. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Socket preservation
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Post-extraction Bone Regeneration
Keywords: tooth extraction; alveolar bone; bone regeneration; laser

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either laser or control group.
Who Masked: Outcomes Assessor
Masking Description: CBCT will be used to assess bone density and the assessors will be unaware of the patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser (Experimental): After extraction, Er:YAG and Nd:YAG lasers used for degranulation, disinfection, deepithelialization, clot stabilization and photobiomodulation.
  Interventions: Device: Er:YAG and Nd:YAG lasers
- Control (Active Comparator): Standard extraction procedure.
  Interventions: Procedure: Standard extraction

INTERVENTIONS:
Device: Er:YAG and Nd:YAG lasers — Extraction followed by Er:YAG laser degranulation, Nd:YAG laser disinfection, Er:YAG deepithelialization, Nd:YAG blood clot stabilization and photobiomodulation. The photobiomodulation step repeated on day 3, 5, and 7.
  Other Names: Twinlight; laser alveolar preservation; LightWalker; Fotona
  Arms: Laser
Procedure: Standard extraction — Standard extraction procedure
  Arms: Control

SUMMARY:
Alveolar bone regeneration after laser-assisted extraction will be compared with bone regeneration after standard extraction procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient requires at least one simple extraction
* Voluntary informed consent to participate in the study

Exclusion Criteria:

* Pregnancy
* Use of photosensitizing medication
* Refuse participation
* Require complicated extraction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change in bone density from immediate post-extraction | 3 months
  Cone Beam Computed Tomography (CBCT)

SECONDARY OUTCOMES:
Bone density | 3 months
  Cone Beam Computed Tomography (CBCT)
Bone thickness | 3 months
  Cone Beam Computed Tomography (CBCT)
Treatment pain | day 1
  On a pain scale from 0 (no pain) to 10 (intolerable pain)
Treatment pain | day 3
  On a pain scale from 0 (no pain) to 10 (intolerable pain)
Treatment pain | day 5
  On a pain scale from 0 (no pain) to 10 (intolerable pain)
Treatment pain | day 7
  On a pain scale from 0 (no pain) to 10 (intolerable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Križaj Dumić, MDD, Principal Investigator — Krizaj d.o.o.
Locations (1):
- Klinika Križaj, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No